CLINICAL TRIAL: NCT06848101
Title: Eye and Carotenoid Augmentation Research and Evaluation (EyeCARE)
Acronym: EyeCARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Daiken Biomedical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB23-0196
Record Dates: First submitted 2025-02-24; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Vision; Eye Health
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carotenoid Complex Supplement (Experimental): 20mg free lutein (10mg/softgel), 4 mg free zeaxanthin (2mg/softgel), 40mg maqui berry extract (20mg/softgel), 6 mg astaxanthin (3 mg/softgel), 80mg bilberry extract (40mg/softgel), flaxseed oil (150mg/softgel), and vitamin E (5IU/softgel)
  Interventions: Dietary Supplement: Carotenoid Group
- Control (Placebo Comparator): flaxseed oil (330mg)
  Interventions: Dietary Supplement: Control (placebo) group

INTERVENTIONS:
Dietary Supplement: Carotenoid Group — Treatment will contain 20mg free lutein (10mg/softgel), 4 mg free zeaxanthin (2mg/softgel), 40mg maqui berry extract (20mg/softgel), 6 mg astaxanthin (3 mg/softgel), 80mg bilberry extract (40mg/softgel), flaxseed oil (150mg/softgel), and vitamin E (5IU/softgel)
  Arms: Carotenoid Complex Supplement
Dietary Supplement: Control (placebo) group — Flaxseed Oil (330mg)
  Arms: Control

SUMMARY:
The primary study outcomes are to investigate the effects of 4-month daily carotenoid complex supplementation on carotenoid status in the macula and skin and visual fatigue among adults 20-45 years of age. Secondary outcomes will examine the supplementation effects on cognitive function.

DETAILED DESCRIPTION:
Lutein and zeaxanthin are carotenoids or plant-based pigments that accumulate in various human tissues including the eye, skin, adipose/fat, and the brain where they play important roles as antioxidants and light filters. Previous correlational work has shown that lutein and zeaxanthin intake is associated with multiple markers of health including visual and cognitive outcomes. However, experimental or intervention research examining the effects of lutein and zeaxanthin supplementation on the accumulation of these carotenoids in the eye and skin and implications for visual and cognitive function is still emerging. Additionally, virtually all the previous research has relied on single nutrient supplementation (e.g., only lutein or zeaxanthin) resulting in limited knowledge of the benefits of providing these carotenoids with other possibly healthful nutrients (e.g., astaxanthin, vitamin E). Accordingly, this project will test the effects of lutein and zeaxanthin supplementation provided in a complex with other antioxidants and nutrients on outcomes of nutritional status in the eye and skin as well as visual and cognitive health. The study aims will be addressed using a double-blind randomized controlled trial design. Adults 20-45 years of age will be asked to participate in a daily 4-month double-blind randomized controlled clinical trial. Treatment group (N=20) participants will be asked to consume 2 daily softgels with a daily total containing 20mg free lutein (10mg/softgel), 4 mg free zeaxanthin (2mg/softgel), 40mg maqui berry extract (20mg/softgel), 6 mg astaxanthin (3 mg/softgel), 80mg bilberry extract (40mg/softgel), flaxseed oil (150mg/softgel), and vitamin E (5IU/softgel). Participants will be asked to consume the supplements with a meal of their choosing. Control group participants will be asked to consume similar-looking placebo softgels over the same period.

ELIGIBILITY:
Inclusion Criteria:

1. not pregnant
2. not breastfeeding
3. absence of hypertension
4. absence of diabetes
5. absence of cerebrovascular disease
6. absence of cardiovascular disease
7. absence of liver disease
8. absence of kidney disease
9. absence of gastrointestinal disease
10. absence of age-related macular degeneration
11. no allergy to carotenoids
12. 20/20 or corrected vision
13. MPOD less than or equal to 0.60
14. Age between 20-45 years

Exclusion Criteria:

1. pregnant
2. breastfeeding
3. presence of hypertension
4. presence of diabetes
5. presence of cerebrovascular disease
6. presence of cardiovascular disease
7. presence of liver disease
8. presence of kidney disease
9. presence of gastrointestinal disease
10. presence of age-related macular degeneration
11. allergy to carotenoids
12. not 20/20 or uncorrected vision
13. MPOD greater than 0.60
14. Younger than 20 years or older than 45 years

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-03-14 (Estimated); Study Completion 2025-03-14 (Estimated)

PRIMARY OUTCOMES:
Macular Pigment Optical Density | From enrollment to end of treatment at 4 months
  Macular carotenoids assessed using heterochromatic flicker photometry

SECONDARY OUTCOMES:
Skin carotenoids | From enrollment to end of treatment at 4 months
  Carotenoids in skin assessed using skin reflection spectroscopy
Visual Fatigue | From enrollment to end of treatment at 4 months
  Visual fatigue as assessed by the Computer Vision Syndrome Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of illinois, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No